CLINICAL TRIAL: NCT04782674
Title: A Prospective Study on the Application of Saliva EBV-DNA Detection in EBV Infection Related Diseases
Brief Title: Study on the Application of Saliva EBV-DNA Detection in EBV Infection Related Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Principal Investigator, Beijing Friendship Hospital
Other Study IDs: saliva EBV-DNA
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: EBV Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Saliva Testing — Saliva EBV-DNA Detection comparing with PBMC and plasma EBV-DNA

SUMMARY:
This study is a single-center, prospective, observational clinical study to evaluate the Application of saliva EBV-DNA Detection in EBV Infection Related Diseases

ELIGIBILITY:
Inclusion Criteria:

1. According to the HLH-04 diagnostic criteria, it meets the HLH diagnostic criteria. EBV infection occurs in cells with EBV-DNA copy number significantly increased in peripheral blood or tissue, or where EBV coding small RNA(EBER) is detected in tissue or peripheral blood. Or Straus' 1988 diagnostic criteria for CAEBV.
2. Informed consent

Exclusion Criteria:

1. Patients who cannot cooperate with saliva collection
2. Patients who are unwilling to cooperate with the project research according to the project research plan.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffer EBV infection related disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Diagnosis | baseline
  The sensitivity and specificity of saliva EBV-DNA detection level as a diagnosis for EBV infection-related diseases, and whether it can replace peripheral blood EBV-DNA monitoring
Monitoring | 2 to 12 weeks after treatment
  The sensitivity and specificity of saliva EBV-DNA detection level as a monitoring method for EBV infection-related diseases, and whether it can replace peripheral blood EBV-DNA monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided